CLINICAL TRIAL: NCT06224504
Title: Combined Mindfulness-Based Stress Reduction and Exercise Intervention for Improving Psychological Well-being in Chinese Patients With Non-Small Cell Lung Cancer
Brief Title: Clinical Effectiveness of Combining Mindfulness-Based Stress Reduction With Exercise Interventione
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Principal Investigator, Wanling Li, Principal Investigator, Shanxi Bethune Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBH-001
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung cancer; Mindfulness-Based Stress Reduction; Exercise intervention; Anxiety; Depression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Anxiety Disorders; Depression | interventions — Mindfulness-Based Stress Reduction; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): routine health education ， psychological nursing， MBSR therapy ， exercise therapy
  Interventions: Behavioral: routine health education; Behavioral: psychological nursing; Behavioral: MBSR therapy; Behavioral: exercise therapy
- the control group (Active Comparator): routine health education ， psychological nursing
  Interventions: Behavioral: routine health education; Behavioral: psychological nursing

INTERVENTIONS:
Behavioral: routine health education — guided the diet of patients, and introduced the knowledge of the disease in detail
Behavioral: psychological nursing — hen the patient has negative emotions, patiently listen to the patient's expression, and timely provide language comfort and guidance to the negative psychological emotions
Behavioral: MBSR therapy — Conducted in small groups once a week for 8 weeks, with each session lasting approximately 1-1.5 hours, encompassed mindfulness-based breathing exercises, dietary interventions, and body scans
  Arms: the intervention group
Behavioral: exercise therapy — Participants were assigned daily tasks for each session, requiring approximately 35-45 minutes per day
  Arms: the intervention group

SUMMARY:
This study is to assess the clinical effectiveness of combining Mindfulness-Based Stress Reduction (MBSR) with exercise intervention in improving anxiety, depression, sleep quality, and mood regulation in Chinese patients with non-small cell lung cancer (NSCLC).The control group received conventional psychological nursing care, while the intervention group received a combination of MBSR and exercise therapy. Pre- and post-treatment scores of anxiety, depression, sleep quality, and the BSRS-5 were compared.

DETAILED DESCRIPTION:
To assess the clinical effectiveness of combining Mindfulness-Based Stress Reduction (MBSR) with exercise intervention in improving anxiety, depression, sleep quality, and mood regulation in Chinese patients with non-small cell lung cancer (NSCLC). A total of 60 lung cancer patients from a hospital in Shanxi Province were selected using convenience sampling and divided into an intervention group and a control group, with 30 patients in each group. The control group received conventional psychological nursing care, while the intervention group received a combination of MBSR and exercise therapy. The two group were evaluated by the questionnaire three times. One day before the intervention, the first questionnaire was conducted, and the basic data of the two groups of patients were collected. The second questionnaire evaluation of anxiety, depression, sleep quality, and the Brief Symptom Rating Scale (BSRS-5) was conducted 6 weeks after the end of the intervention, and the third questionnaire evaluation was conducted 8 weeks after the end of the intervention to evaluate the intervention effect of the two groups. Pre- and post-treatment scores of anxiety, depression, sleep quality, and the BSRS-5 were compared.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with non-small cell lung cancer
* patients aged between 20 and 74 years, without gender limitation
* a score of 4-14 on the Short Symptom Rating Scale (BSRS-5)
* a clinical prognosis of at least 6 months
* clear consciousness, good functional ability, and unrestricted language communication
* written informed consent provided by the patient

Exclusion Criteria:

* patients with severe physical illnesses or symptoms that impede learning and are considered life-threatening
* patients with a BSRS-5 assessment score > 15 and suicidal ideation > 2
* patients unable to accurately describe their symptoms
* patients with limited cooperation ability
* patients who have previously undergone MBSR or other positive-thinking-focused psychotherapy methods

Ages: 44 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
SAS score | one day before the intervention
  Self-Rating Anxiety Scale (SAS)
SAS score | at 6 weeks after the intervention
  Self-Rating Anxiety Scale (SAS)
SAS score | at 8 weeks after the intervention
  Self-Rating Anxiety Scale (SAS)
SDS score | one day before the intervention
  Self-Rating Depression Scale (SDS)
SDS score | at 6 weeks after the intervention
  Self-Rating Depression Scale (SDS)
SDS score | at 8 weeks after the intervention
  Self-Rating Depression Scale (SDS)
BSRS-5 score | one day before the intervention
  the five-item Brief Symptom Rating Scale (BSRS-5)
BSRS-5 score | at 6 weeks after the intervention
  the five-item Brief Symptom Rating Scale (BSRS-5)
BSRS-5 score | at 8 weeks after the intervention
  the five-item Brief Symptom Rating Scale (BSRS-5)
PSQI score | one day before the intervention
  Pittsburgh Sleep Quality Index (PSQI)
PSQI score | at 6 weeks after the intervention
  Pittsburgh Sleep Quality Index (PSQI)
PSQI score | at 8 weeks after the intervention
  Pittsburgh Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Wanling Li, Principal Investigator — Shanxi Bethune Hospital
Locations (1):
- Combined Mindfulness-Based Stress Reduction and Exercise Intervention for Improving Psychological Well-being in Chinese Patients with Non-Small Cell Lung Cancer, Taiyuan, Shanxi, China